CLINICAL TRIAL: NCT02545101
Title: A Non Interventional, Retrospective Study on Real World Usage and Treatment Outcomes of Patients Treated With Tolvaptan for Hyponatraemia Due to the SIADH.
Brief Title: An Observational Study on Real-world Use and Outcomes of Patients Treated With Tolvaptan for Hyponatraemia Due to SIADH
Acronym: SAMPLE
Status: Completed | Type: Observational
Sponsor: Otsuka Pharmaceutical Europe Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 156-303-00034
Record Dates: First submitted 2015-09-07; First posted 2015-09-09 (Estimated); Results first posted 2018-02-05 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-02

CONDITIONS: Hyponatremia; Syndrome of Inappropriate ADH (SIADH) Secretion
Keywords: Hyponatremia due to SIADH; tolvaptan
MeSH Terms: conditions — Hyponatremia; Inappropriate ADH Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective chart review non-interventional study designed to collect real world data on the use and outcomes of tolvaptan for the treatment of patients with hyponatraemia secondary to syndrome of inappropriate antidiuretic hormone (SIADH) secretion.

ELIGIBILITY:
Inclusion Criteria:

* Provision of patient informed consent unless a) not required by local regulations, b) it would take a non reasonable effort or c) if the source patient is deceased or untraceable.
* Female and/or male patients aged 18 years and over.
* Patients who received at least 2 doses of tolvaptan, for the treatment of one occurrence of hyponatraemia secondary to SIADH.

Exclusion Criteria:

* A patient cannot take part in this study if participating in any other clinical study in which the medicinal product aims to treat the causes or symptoms of hyponatraemia at the time of the hyponatraemia episode being documented in the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients are ≥ 18 years old and have been treated with at least 2 doses of tolvaptan for one occurrence of hyponatraemia secondary to SIADH during 2014. If the number of patients treated with tolvaptan in 2014 in the participating centres is not sufficient to reach the intended sample size, this retrospective enrolment period could be extended to include patients treated in 2013.
  A mix of centres and treating departments (e.g. endocrinology, nephrology, etc.), will be selected within each participating country in order to provide a sufficiently representative sample of patients treated with tolvaptan for hyponatraemia secondary to SIADH.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Department, Study Director — Otsuka Europe
Locations (7):
- Germany (4):
  - Bochum
  - Chemnitz
  - Dresden
  - Lübeck
- Spain (3):
  - Córdoba
  - Madrid
  - Santiago de Compostela

REFERENCES:
- [Derived] Pose-Reino A, Runkle de la Vega I, de Jong-Laird A, Kabra M, Lindner U. Real-World, Non-Interventional, Retrospective Study (SAMPLE) of Tolvaptan in Patients with Hyponatraemia Secondary to the Syndrome of Inappropriate Antidiuretic Hormone Secretion. Adv Ther. 2021 Feb;38(2):1055-1067. doi: 10.1007/s12325-020-01560-2. Epub 2020 Dec 11. PMID 33306187

RESULTS

PARTICIPANT FLOW:
Groups:
- Tolvaptan: Adult patients who received at least 2 doses of tolvaptan for the treatment of one occurrence of hyponatraemia secondary to SIADH.
Period: Overall Study
Arm/Group | Tolvaptan
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tolvaptan
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.9 (14.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 47
Region of Enrollment [Number; unit: participants]
  Germany | 44
  Spain | 56
Weight [Mean (Standard Deviation); unit: kg] — Population: number of patients meeting the criterion
  kg
    number analyzed (Participants) | 89
    (all) | 68.8 (15.03)
Height [Mean (Standard Deviation); unit: meters] — Population: number of patients meeting the criterion
  meters
    number analyzed (Participants) | 89
    (all) | 1.632 (0.0831)
Body Mass Index [Mean (Standard Deviation); unit: Kg/m^2] — Population: number of patients meeting the criterion.
  Kg/m^2
    number analyzed (Participants) | 89
    (all) | 25.781 (5.2890)

OUTCOME MEASURES:

1. Primary Outcome: Change in Sodium Levels From Start of Treatment With Tolvaptan Until Hospital Discharge
Description: The primary variable of the study was the change in sodium levels from baseline to discharge or the final available measurement for patients who were not discharged (up to 6 weeks after treatment initiation).
Time Frame: From Baseline Up to discharge (or a maximum of 6 weeks after start of treatment)
Population: Baseline sodium level was not available for 4 patients
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tolvaptan
Number analyzed (Participants) | 96
mmol/L | 10.3 (6.42)

2. Secondary Outcome: Change in Sodium Levels 24 Hours After Treatment Initiation
Description: Change in sodium level from last value prior to receiving tolvaptan until last available measurement within 24 hours of initiation of tolvaptan
Time Frame: From Baseline (treatment initiation with tolvaptan) up to 24 hours afterwards
Population: Only patients with a value at both baseline and 24 hours of initiation of tovaptan were included in the change from baseline
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tolvaptan
Number analyzed (Participants) | 95
mmol/L | 3.3 (4.53)

3. Secondary Outcome: Change in Sodium Levels 6 Weeks After Treatment Initiation
Description: Change in sodium level from last value prior to receiving tolvaptan until last available measurement up to week 6
Time Frame: From Baseline (treatment initiation with tolvaptan) up to 6 weeks afterwards
Population: only patients with a value at both baseline and that time point are included in the change
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tolvaptan
Number analyzed (Participants) | 96
mmol/L | 11.8 (6.45)

4. Secondary Outcome: Time (Hours) to Sodium Normalisation
Description: Time (hours) to sodium normalisation, defined as a serum sodium level > 135 mmol/L, by evaluation of serum sodium levels in relation to the episode of hyponatraemia secondary to SIADH being captured in the study (up to 6 weeks after treatment initiation).
Time Frame: From Baseline (treatment initiation with tolvaptan) up to 6 weeks afterwards
Population: Exact time was available for 64 patients, so the analysis "in hours" had a n=64
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Tolvaptan
Number analyzed (Participants) | 64
hours | 115.5 [72 to 187]

5. Secondary Outcome: Percentage of Participants Distributed by the Primary Disease Diagnoses Leading to SIADH (Cancer, Pulmonary Disease, CNS Disorder, Etc.,)
Description: Primary disease diagnoses leading to SIADH by evaluation of diagnosis information in relation to the episode of hyponatraemia being captured in the study from the patient's medical records
Time Frame: Baseline
Measure: Number; unit: % of participants
Arm/Group | Tolvaptan
Number analyzed (Participants) | 100
% of participants
  Cancer | 27
  Medication | 20
  CNS disorder | 11
  Pulmonary disease | 7
  Hereditary causes | 3
  Other (mainly unknown/idiopathic origin) | 32

6. Secondary Outcome: Symptoms Associated With Hyponatraemia (Number of Symptomatic/Asymptomatic Patients in the Study Population)
Description: symptoms associated with hyponatraemia by evaluation of symptomatology information in relation to the episode of hyponatraemia being captured in the study from the patient's medical records
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Tolvaptan
Number analyzed (Participants) | 100
Participants | 83

7. Secondary Outcome: Percentage of Participants Distributed by the Specialties of Their Clinicians Prescribing Tolvaptan (e.g., Endocrinologists, Nephrologists, Oncologists, Etc.,)
Description: specialty of the clinician prescribing tolvaptan by evaluation of details of the physician who prescribed tolvaptan for the episode of hyponatraemia being captured in the study from the patient's medical records
Time Frame: Baseline
Measure: Number; unit: % of participants
Arm/Group | Tolvaptan
Number analyzed (Participants) | 100
% of participants
  Endocrinology | 40
  Nephrology | 25
  Internal medicine | 19
  Emergency Room Dept | 6
  Oncology | 5
  Other | 5

8. Secondary Outcome: Average Daily Dose of Tolvaptan Used and Treatment Duration (Expressed in Days) for the Episode of Hyponatraemia Being Captured in the Study
Description: Average daily dose of tolvaptan used and treatment duration (expressed in days) for the episode of hyponatraemia secondary to SIADH being captured in the study by evaluation of dosing information (and dates) from the patient's medical records (up to 6 weeks after the initiation of tolvaptan treatment).
  For these outcome measures, only days on treatment were considered (e.g. if tolvaptan treatment was interrupted and resumed afterwards, the days withot treatment were not considered).
Time Frame: From Baseline (treatment initiation with tolvaptan) up to 6 weeks afterwards
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Tolvaptan
Number analyzed (Participants) | 100
mg | 12.67 (9.173)

9. Secondary Outcome: Time (Days) to Sodium Normalisation
Description: Time (days) to sodium normalisation, defined as a serum sodium level > 135 mmol/L, by evaluation of serum sodium levels in relation to the episode of hyponatraemia secondary to SIADH being captured in the study (up to 6 weeks after treatment initiation).
Time Frame: From Baseline (treatment initiation with tolvaptan) up to 6 weeks afterwards
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Tolvaptan
Number analyzed (Participants) | 100
days | 7 [5 to 10]

10. Other Pre Specified Outcome: Concomitant Treatments to Tolvaptan (Number and Percentage of Subjects Taking Concomitant Medications Will be Summarized by Anatomical Therapeutic Chemical (ATC) Classification)
Description: Only medications taken by more than 5% of the study population are presented
Time Frame: From baseline (tolvaptan treatment initiation) up to 6 weeks after treatment initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Tolvaptan
Number analyzed (Participants) | 100
Participants
  Acetylsalicylic acid | 27
  Omeprazole | 25
  Amlodipine | 23
  Ramipril | 18
  Dexomethasone | 15
  Pantoprazole | 15
  Enoxaparin | 14
  Lorazepam | 14
  Metamizole | 13
  Simvastatin | 13
  Acetominophen | 11
  Levothyroxine | 10
  Metformin | 10
  Enalapril | 10
  Torasemide | 8
  Ondansetron | 8
  Fursosemide | 7
  Insulin | 7
  Levetiracetam | 7
  Lactulose | 7
  Atorvastatin | 7
  Metoprolol succinate | 7
  Metoclopramide | 7
  Bisoprolol | 6
  Metoprolol | 6
  Normal saline | 6
  Salbutamol | 6

11. Post Hoc Outcome: Time (Days) to Hospital Discharge up to 6 Weeks After Treatment Start
Time Frame: From Baseline (treatment initiation with tolvaptan) up to 6 weeks afterwards
Population: Originally, the idea was to analyse this out come in "hours", but due to missing data, it was also analysed in "days".
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Tolvaptan
Number analyzed (Participants) | 100
days | 7.0 [6.0 to 9.0]

12. Secondary Outcome: Number of Participants With Presence of Different Symptoms Associated With Hyponatraemia
Description: as for outcome 6
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Tolvaptan
Number analyzed (Participants) | 100
Participants
  lethargy | 41
  gait disorder | 37
  nausea | 33
  disorientation | 31
  drowsiness | 30
  anorexia | 28
  confusion | 28
  vomiting | 24
  restlessness | 15
  brain damage | 10
  headache | 10

13. Secondary Outcome: Average Treatment Duration for the Episode of Hyponatraemia Being Captured in the Study
Description: Average treatment duration for the episode of hyponatraemia secondary to SIADH being captured in the study by evaluation of dosing information (and dates) from the patient's medical records (up to 6 weeks after the initiation of tolvaptan treatment).
  For these outcome measures, only days on treatment were considered (e.g. if tolvaptan treatment was interrupted and resumed afterwards, the days withot treatment were not considered).
Time Frame: From Baseline (treatment initiation with tolvaptan) up to 6 weeks afterwards
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tolvaptan
Number analyzed (Participants) | 100
days | 27.96 (16.479)

14. Other Pre Specified Outcome: Prior Treatments Before Tolvaptan (Number and Percentage of Subjects Taking Prior Medications Will be Summarized by Anatomical Therapeutic Chemical (ATC) Classification)
Description: Only medications taken by more than 5% of the study population are presented
Time Frame: From 12 months up to baseline (tolvaptan treatment initiation)
Measure: Count of Participants; unit: Participants
Arm/Group | Tolvaptan
Number analyzed (Participants) | 100
Participants
  Furosemide | 10
  Levofloxavin | 7
  Normal Saline | 6

ADVERSE EVENTS:
Time Frame: Study period was defined for each patient as: from start of tolvaptan treatment until 6 weeks afterwards maximum.
Description: Treatment-emergent adverse event defined as adverse event (AEs) that started or worsened after the start of the administration of tolvaptan, i.e. meaning temporal association but not necessarily causality/relationship (investigators were not asked about this).
  Please note that collection of AE, as the study itself, was retrospective.
Arm/Group | Tolvaptan
All-Cause Mortality (participants affected / at risk) | 3/100
Serious Adverse Events (participants affected / at risk) | 10/100
Other Adverse Events (participants affected / at risk) | 12/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tolvaptan (N=100)
WOUND INFECTION (Infections and infestations) | 1 (1) — INFECTION OF OPEN FRACTURES
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) — HYPONATREMIA EPISODE
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
DEATH (General disorders) | 1 (1) — NATURAL DEATH (EXTREMELY OLD DEATH)
BLOOD SODIUM INCREASED (Investigations) | 1 (1) — RAPID RAISE IN SODIUM LEVELS
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) — NEUTROPENIA POST-CHEMOTHERAPY
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Fatal for 1 patient.
EPILEPSY (Nervous system disorders) | 1 (1) — EPILEPTIC SEIZURE
SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — EXITUS BY SMALL CELL LUNG CANCER
SYNCOPE (Nervous system disorders) | 1 (1)
MENINGITIS (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tolvaptan (N=100)
THIRST (General disorders) | 1 (1)
EAR INFECTION (Infections and infestations) | 1 (1) — OTITIS
ORAL CANDIDIASIS (Infections and infestations) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 1 (1)
CHOLANGITIS ACUTE (Hepatobiliary disorders) | 1 (1) — ACUTE COLANGITIS WITH FEVER AND ELEVATION OF LIVER ENZYMES
BLOOD SODIUM DECREASED (Investigations) | 1 (1)
BLOOD SODIUM ABNORMAL (Investigations) | 1 (1) — NO IMPROVE SODIUM LEVELS
DIARRHOEA (Gastrointestinal disorders) | 1 (1)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1)
BLOOD SODIUM INCREASED (Investigations) | 2 (2)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1)
SEIZURE (Nervous system disorders) | 1 (1)
CYSTITIS (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
As a multicentre study, the first publication shall be based on consolidated analysed data from all centres, i.e. the publication of results from individual institution/Investigator is not allowed before the publication of the full study results.

The PI agrees to give the sponsor 60 days to review the communications. If case of propietary information inadvertenly divulged, intellectual property rights at risk or inaccurate information presented, changes can be required by the sponsor.